CLINICAL TRIAL: NCT05933174
Title: Promoting Alternatives to Sulfonylureas to Improve Patient Safety in Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ian J. Neeland, MD (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Ian J. Neeland, MD, Principal Investigator, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20230836; Neeland AHA 23SCISA1144816 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Type2diabetes
Keywords: Sulfonylureas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prompt-sheet (Experimental): Question-prompt group patients will receive a simple prompt sheet with the questions with which they will encouraged to use to guide a conversation with their provider at their next visit for routine diabetes care. These questions are based on recommendations from the Agency for Healthcare Research and Quality's Question Builder App and also on recommendations from the Canadian Deprescribing Network which specifically addresses SU use.
  Interventions: Other: Prompt-sheet
- Usual education (Active Comparator): Control group patients will be sent an information brochure with content from the NIDDK about diabetes medications (https://www.niddk.nih.gov/health-information/diabetes/overview/insulin-medicines-treatments).
  Interventions: Other: Usual education

INTERVENTIONS:
Other: Prompt-sheet — Simple prompt sheet with which participants will encouraged to use to guide a conversation with their provider at their next visit for routine diabetes care. These questions are based on recommendations from the Agency for Healthcare Research and Quality's Question Builder App and also on recommendations from the Canadian Deprescribing Network which specifically addresses SU use.
  Arms: Prompt-sheet
Other: Usual education — Control group patients will be sent an information brochure with content from the NIDDK about diabetes medications (https://www.niddk.nih.gov/health-information/diabetes/overview/insulin-medicines-treatments).
  Arms: Usual education

SUMMARY:
Sulfonylurea medications are unsafe for older patients with diabetes. They are associated not only with hypoglycemia, but also with falls and increased cardiovascular risk. Yet they continue to be prescribed frequently. Indeed, older adults with type 2 diabetes, who are especially prone to adverse effects, are more likely to be prescribed sulfonylureas than younger patients. This is unfortunate since over the past several years, newer, safer, and more effective classes of medications (GLP-1 agonists and SGLT2-inhibitors) have emerged. The investigators acknowledge that sulfonylureas are inexpensive and that their low cost is a driver of continued use. However, the investigators believe patients and providers should have discussions about the risks of sulfonylureas and safer and more effective alternatives, to make diabetes care safer overall in ambulatory settings. Our research is designed to promote such discussions. The investigators will first identify patients taking sulfonylureas regularly. Next, using recommendations from AHRQ and the Canadian Deprescribing Network, the investigators will empower patients to discuss their medications with their providers through a simple question prompt sheet. Patients will be divided into an intervention group which receives explicit prompting questions, and a control group that receives a general brochure on diabetes medications. Health care providers will receive education about newer diabetes medications through case-based discussions and academic detailing. Finally the investigators will measure key outcomes including the proportion of patients who have discussions about sulfonylureas and alternatives, rates of discontinuation, and measures of control of diabetes and associated cardiovascular risks. The investigators will also evaluate the experiences of patients and providers qualitatively through brief, semi-structured interviews. Should our multi-faceted, patient-oriented intervention prove effective in promoting discussions of sulfonylureas and alternatives, and also discontinuation of sulfonylureas and switching to newer alternatives, the investigators will incorporate our prompting questions into routine care for patients taking sulfonylureas. Our intervention can be easily disseminated to other settings and therefore has considerable potential to improve safety among patients with type 2 diabetes nationwide.

DETAILED DESCRIPTION:
The objectives of this study are to systematically (a) identify middle-aged and older adults taking SU within a large integrated health system, and empower them to explore alternative, evidence-based treatments with their primary care providers to address and implement the ADA practice guideline as an actionable target to improve patient safety; and (b) engage our primary care providers in a systematic quality implementation and improvement program that includes education about contemporary T2D guideline recommendations, benefits, and drawbacks of different classes of agents, and formulary alternatives to SU. These objectives will be accomplished in the following 3 aims:

1. Empower patients to discuss treatments options with their primary care provider.

   Using an electronic data warehouse, the investigators will identify patients aged ≥45 years with type 2 diabetes who are currently prescribed SU and implement a strategy to encourage patients to discuss SU and alternatives with their primary care providers using a question-based prompt sheet. A control group will receive an overview sheet of diabetes medications.
2. Engage primary care providers in a quality implementation and improvement program.

   The program includes education about contemporary T2D guideline recommendations, benefits, and drawbacks of different classes of agents, and formulary alternatives to SU. An academic detailer will visit each primary care practice up to twice during the study period to provide targeted education about alternatives to SU to promote safety.
3. Measure key process outcomes and patient-centered outcomes at regular intervals.

Participants will be surveyed every 3 months during their first year of participation to identify if they had discussed alternatives. The investigators hypothesize that half of intervention group patients will have had such discussions compared with only 25% in the control group. Other outcomes will include assessment of hypoglycemia symptoms, discontinuation rates of SU, initiation of new medications, diabetes and financial distress (via surveys), and clinical outcomes (extracted from the electronic medical record) including glycosylated hemoglobin (Hb A1c), body weight, blood pressure, and lipids.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Type 2 diabetes (diagnosed on or before 12/31/2021)
* Current/active prescription for one or more SU medications
* Established care (≥2 visits) with UH primary care provider (PCP) since 2021

Exclusion Criteria:

* Type 1 diabetes
* PCP provides a reason why patient participation is inappropriate (e.g., known cost barriers without any alternatives, prior discussion with patient about alternatives, etc.)
* Patient unable or unwilling to have conversation with their PCP regarding SU
* Unable to provide informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified gender
Enrollment: 220 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who had a conversation with their primary care provider about SU use and alternatives for their diabetes management | 12 months
  Proportion of patients who had a conversation with their primary care provider about SU use and alternatives for their diabetes management

SECONDARY OUTCOMES:
Proportion of patients who switched from a SU to an alternative medication | 12 months
  Proportion of patients who switched from a SU to an alternative medication
Proportion of patients who discontinued a SU | 12 months
  Proportion of patients who discontinued a SU
Proportion of patients who experienced a hypoglycemia event by self-report | 12 months
  Proportion of patients who experienced a hypoglycemia event by self-report
Hb A1c | 12 months
  glycosylated hemoglobin
BMI | 12 months
  body mass index
Blood pressure (systolic and diastolic) | 12 months
  Blood pressure (systolic and diastolic)
Lipid levels | 12 months
  Lipid levels
The Personal Financial Well-being Scale | 12 months
  . The financial well-being scale is a free tool to help measure the financial well-being of people you serve. The scale, which was developed and rigorously tested by The Consumer Financial Protection Bureau, contains 10 questions to capture how people feel about their financial security and freedom of choice, plus 2 questions to assist with scoring. Responses to the questions can be converted into an overall financial well-being "score" between 0 and 100.
Diabetes Distress Scale | 12 months
  17-item self-report survey to assess an individual's level of stress related to living with diabetes. Each question has an answer rating from 1 ("not a problem") to 5 ("a very serious problem").

CONTACTS AND LOCATIONS:
Overall Officials: Ian Neeland, MD, Principal Investigator — University Hospital Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No